CLINICAL TRIAL: NCT05590338
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamic of a Single Intravenous Dose of GSK1070806 Administered to Healthy Male and Female Caucasian, Chinese and Japanese Participants Aged 18 to 65 Years of Age Inclusive
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic of GSK1070806 After a Single Intravenous Dose in Healthy Male and Female Caucasian, Chinese and Japanese Participants Aged 18 to 65 Years of Age Inclusive
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 218841
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Dermatitis, Atopic
Keywords: Immunoglobulin G1 (IgG1) antibody; Interleukin-18 (IL-18); GSK1070806; 218841
MeSH Terms: conditions — Dermatitis, Atopic | interventions — GSK1070806

STUDY DESIGN:
Intervention Model Description: In Part A the participants will be randomly assigned in each arm to receive either active or placebo interventions.
  In Part B the participants will be assigned to receive only active intervention.
Who Masked: Participant, Investigator
Masking Description: In Part A the participants and investigators will be masked. In Part B there will be no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: GSK1070806 (Experimental): Participants in Part A will receive single dose of GSK1070806 intravenous (IV) infusion
  Interventions: Drug: GSK1070806
- Part B: GSK1070806 (Experimental): Participants in Part B will receive single dose of GSK1070806 IV bolus
  Interventions: Drug: GSK1070806
- Part A: Placebo (Placebo Comparator): Participants in Part A will receive single dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1070806 — Participants will receive GSK1070806
  Arms: Part A: GSK1070806; Part B: GSK1070806
Drug: Placebo — Participants will receive placebo
  Arms: Part A: Placebo

SUMMARY:
This study is divided into two parts:

Part A of the study is double blinded, randomized, placebo-controlled and aims to assess the safety, tolerability, pharmacokinetics (PK) and Pharmacodynamic (PD) effect of a single intravenous (IV) infusion dose of GSK1070806 when administered to healthy participants of Japanese, Chinese and European/Caucasian ancestry.

Part B of the study is an open label single cohort arm to assess the safety, tolerability, PK and PD effect of a single IV bolus low dose of GSK1070806 in healthy participants of European/Caucasian ancestry.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring [12-lead Electrocardiogram (ECGs)]
* Between 18 and 65 years of age inclusive, at the time of signing the informed consent
* Body weight within the range 45 - 100 kilograms (kg) and body mass index (BMI) within the range 18-32 kilogram/meter square (kg/m^2) (inclusive)
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:
* Is a woman of non-childbearing potential (WONCBP) OR
* Is a woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective [with a failure rate of less than 1 percent (<1%) per year], with low user dependency
* Capable of giving signed informed consent
* Participants of Japanese ancestry are eligible based on meeting all of the following:
* Healthy male and female participants born in Japan
* Descendants of four ethnic Japanese grandparents and two ethnic Japanese parents
* Have lived outside Japan for less than 10 years at the time of screening
* Chinese participants are eligible based on meeting all of the following:
* Healthy male and female participants born in mainland China, Hong Kong, Macau or Taiwan
* Descendants of four ethnic Chinese grandparents and two ethnic Chinese parents
* Have lived outside mainland China, Hong Kong, Macau or Taiwan for less than 10 years at the time of screening
* Participants of Caucasian/European ancestry are eligible if they self-identify to be of Caucasian/European ancestry and have 2 parents of Caucasian/European ancestry and 4 grandparents of Caucasian/European ancestry

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, immunological, metabolic, musculoskeletal or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data
* Personal or family history of cardiomyopathy
* Known varicella, herpes zoster, or other severe viral infection within 6 weeks of anticipated dosing on Day 1. Or history of recurrent herpes reactivation in the past 2 years
* Evidence of active or latent tuberculosis (TB) as documented by medical history, examination, and TB testing with a positive (not indeterminate) QuantiFERON test
* History or evidence of clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, anaphylaxis, erythema multiforme major, linear immunoglobulin A (IgA) dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis)
* Lymphoma, leukemia, or any malignancy except for basal cell carcinomas of the skin that have been resected with no evidence of metastatic disease for 5 years
* Alanine transaminase (ALT) greater than (>) 1.5x upper limit of normal (ULN)
* Total bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or previous uncomplicated cholecystectomy more than 3 months ago)
* Corrected QT using Bazett's formula (QTcB) (Bazett) or Corrected QT using Fridericia's formula (QTcF) (Fridericia) interval >450 milli second (msec)
* History of Stevens Johnson Syndrome
* Known immunodeficiency
* Previous or current history of bleeding diathesis
* Intended use of over the counter or prescription medication including herbal medications within 7 days (or 14 days if the drug is a potential enzyme inducer) or five half-lives (whichever is longer) prior to dosing until final follow-up visit
* Live vaccine(s) or plans to receive such vaccines within 2 months of dosing until final follow-up visit
* Participation in the study would result in loss of blood or blood products in excess of 500 milli liter (mL) within 3 months
* Current enrollment or past participation in any other clinical study involving an investigational study intervention or any other type of medical research within the last 30 days, 5 half-lives or twice the duration of the known pharmacological/biological effect from the last dosing before dosing day in the current study
* Coronavirus strain 19 (COVID-19) (severe acute respiratory syndrome - Coronavirus-2 (SARS CoV-2)):
* Has had COVID-19 infection within 4 weeks of the initial screening visit
* Positive coronavirus test (COVID-19: SARS-CoV-2 Polymerase chain reaction (PCR) or rapid antigen test) at initial screening
* Signs and symptoms suggestive of COVID-19 (i.e., fever, cough, etc.) within 14 days of initial screening Known COVID-19-positive contacts within 14 days of initial Screening, at any time during the Screening Period, or within 14 days of dosing on Day 1
* Active substance abuse or a history of substance abuse within 6 months prior to the initial Screening visit. Substance abuse including cannabis is also prohibited during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Part A: Serum GSK1070806 area under the concentration-time curve from time zero extrapolated to infinity (AUC[0-∞]) | Up to Week 24
Part A: Serum GSK1070806 area under the concentration-time curve from time zero to the last quantifiable time (AUC(0-t)) | Up to Week 24
Part A: Maximum observed serum concentration (Cmax) of GSK1070806 | Up to Week 24
Part A: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to Week 24

SECONDARY OUTCOMES:
Part B: Number of participants with AEs and SAEs | Up to Week 32
Part A: Total IL-18 concentrations in serum | Up to Week 24
Part B: Total IL-18 concentrations in serum | Up to Week 32
Part A: Number of participants with anti-drug antibody (ADA) formation | Up to Week 24
Part B: Number of participants with ADA formation | Up to Week 32

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - GSK Investigational Site, Cypress, California
  - GSK Investigational Site, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/